CLINICAL TRIAL: NCT06754163
Title: Pilot Study Designed in a Phase IV Clinical Trial Framework: Evaluating the Effect of the STEP@STAH Semaglutide Protocol on the Physical Health Measures of Atypical Antipsychotic-Treated Patients in a Secure Mental Healthcare Setting
Brief Title: Evaluating the Effect of the STEP@STAH Semaglutide Protocol on the Physical Health Measures of Atypical Antipsychotic-Treated Patients
Acronym: STEP@STAH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St Andrew's Healthcare (Other)
Collaborators: Loughborough University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024/254
Record Dates: First submitted 2024-12-17; First posted 2024-12-31 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Obesity and Obesity-related Medical Conditions; Psychiatric Disorders
Keywords: semaglutide; wegovy; GLP-1 agonist
MeSH Terms: conditions — Obesity; Mental Disorders | interventions — semaglutide; Diet; Exercise

STUDY DESIGN:
Intervention Model Description: Wegovy is the medication that will be used in the trial. The dosage schedule is available in the summary of product characteristics with a maintenance dose of 2.4 mg or to the maximum tolerated dose. The non-medication component of the intervention will be coordinated by the Occupational Therapy Technical Instructors (OT TIs). Staff will be provided with an information sheet which will emphasise the importance of a multi-disciplinary approach of the 2-year study period. Key points to be highlighted include:
  * Encourage patients to increase their physical activity
  * Remind patients to reduce their daily calorie intake
  * Encourage and support patients to diligently record their physical activity and dietary intake on their Food/Activity/Sleep (FAS) Diary Sheets This coordinated effort aims to support patients effectively and ensure the success of the study through consistent and comprehensive care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evaluating the Effect of the STEP Protocol on Physical Health Measures (Experimental): The primary aim of the study is to assess the impact of treatment with semaglutide, in combination with a healthy lifestyle (including diet and exercise) on the physical health measures of patients in St Andrew's who have atypical antipsychotic induced weight gain. There is significant evidence that atypical antipsychotic drugs (olanzapine and clozapine) can cause patients to put on weight, partly by increasing their appetite. A significant number of people on this class of drugs are considered as overweight or obese. However, no studies have been carried out to determine whether weight loss-associated drugs such as semaglutide, in association with a healthy lifestyle, may be able to overcome this problem. Although semaglutide has been shown to be effective in the general population, this may be more complex in this group of people as it may interact with the anti-psychotic drugs which may prevent it from acting effectively.
  Interventions: Drug: Semaglutide in combination with a healthy lifestyle intervention (diet and exercise)

INTERVENTIONS:
Drug: Semaglutide in combination with a healthy lifestyle intervention (diet and exercise) — Wegovy (semaglutide) will be provided as an induction dose of 0.25 mg, titrated up every 4 weeks to 0.5 mg, 1.0 mg, 1.7 mg and 2.4 mg, will be given, with a maintenance dose of 2.4 mg or to the maximum tolerated dose.
  To reduce the likelihood of gastrointestinal symptoms, the dose should be escalated over a 16-week period to a maintenance dose of 2.4 mg once weekly. The semaglutide injection will be administered once weekly on the same day of the week throughout the study period. Injections will be administered in the thigh, abdomen or upper arm at any time of the day. As part of the multi-disciplinary approach taken in the STEP trials of Wegovy, patients willl be encouraged to
  * Increase their physical activity
  * Reduce their daily calorie intake
  * Record their physical activity and dietary intake on their Food/Activity/Sleep (FAS) Diary Sheets A secondary goal is to achieve sustained improvements in participants' activity levels and awareness of a healthy diet.

SUMMARY:
A significant number of patients who are prescribed anti-psychotic medication such as clozapine are considered as clinically obese (BMI >35.0). While this may be associated with the appetite promoting properties of the drug, other factors including apathy and lack of physical activity and exercise can exacerbate the weight gain. For those patients who are in a secure care setting and who have restrictions on movement, this provides a particular challenge.

Therefore, a pharmacological option to assist in promoting weight loss would be an attractive option for patients who have reached levels of obesity and for whom diet and exercise alone may not be sufficient. The GLP-1 agonist class of drugs, including semaglutide (Wegovy®), have been approved for the treatment of patients as an adjunct to diet and exercise and for weight loss in adults who have a BMI of 30 kg/m² or greater (obese) or weight-related health problems. The aim of this study is to determine whether long-term treatment with Semaglutide (Wegovy®), in combination with dietary advice, exercise and psychological support, will decrease the weight gain associated with anti-psychotic treatment. Patients will be chosen for the trial according to NICE guidelines for referral to a weight management plan. In addition to the weekly Semaglutide (Wegovy®) injection, they will have regular access to dietary and exercise support as part of an overall healthy lifestyle plan which will form part of their overall care plan. They will also be provided with psychological support as a previous trial demonstrated that behavioural support was important, especially at the early stages of such therapy. The patients' progress will be monitored (weight, activity, diet) throughout the duration of the trial. The results will identify those patients who are most likely to benefit from this therapy and can be used to generate treatment guidelines."

DETAILED DESCRIPTION:
The purpose of the study is to determine whether patients who have gained weight due to being prescribed anti- psychotic drugs (olanzapine or clozapine) and have become clinically obese (BMI>35.0) will react to the GLP-1 agonist class of drugs, including semaglutide (Wegovy®), which have been authorised for the treatment of patients as an adjunct to diet and exercise and for weight loss. These have been demonstrated to be effective in adults who are obese due to general overeating and lack of exercise (general lifestyle factors). However, there have been no studies carried out on patients who have had drug-induced weight gain where the drugs have had their impact, at least in part, by altering the body's metabolism. However, weight gain for patients who are treated with anti-psychotic medication is a complex issue as it cannot be solely ascribed to the drugs, as these people tend to be less active and by default to be more immobile. Therefore, the aim of this study is to determine whether GLP-1 agonists (and specifically semaglutide), in combination with dietary and exercise advice (the "NEW You" healthy lifestyle programme) will have a similar impact to those who are obese due to an unhealthy lifestyle which is not drug-induced. Patients are acutely aware of the impact of anti-psychotic medication on their weight and have discussed options with their clinicians.

However, they realise that exercise alone is not sufficient, and that certain drugs increase appetite. Therefore, informal discussions have led to a discussion on the potential use of medication which may assist in weight loss in conjunction with an overall healthy lifestyle (diet and exercise). This was part of the impetus to develop the trial initially at St Andrew's. However, in order to ensure that the evidence generated was robust, it was decided that it should be in the form of a phase 4 observational trial with specific outcome measures. As it would not be feasible to have a placebo control group, it will be in the form of a pre-post analysis.

Recruitment:

Patients who are eligible to enrol in the trial will be identified by their responsible clinician. They will then be approached by a member of the research team who will explain the trial, what it involves and the potential benefits. In particular, they will be made aware that the programme is not just a drug trial but will also involve engagement in a healthy lifestyle programme where the participants will be encouraged to become aware of their diet and also to engage in exercise. Expert members of the multidisciplinary team will provide support throughout the trial and the participants will be made aware of this through the research team. The trial will also be an integral part of their care plan.

Consent:

Patients should be deemed by their responsible clinician as being capable of giving consent to participate in the study and to engage in the interventions such as keeping a food, exercise and sleep diary with the assistance of a staff member.

Risks, burdens and benefits:

As Wegovy is a routinely available drug that will be prescribed under NICE guidelines with patients and staff being made aware of the potential side effects, the risks will be minimal. Full information about the trial will be available in the patient information sheet and support information will be available in the NEW You healthy lifestyle programme documentation which was developed at St Andrew's in 2020 as part of an NHS Commissioning and Quality Innovation (CQUIN) Framework with significant patient input. Participation in the study should result in an overall healthier lifestyle with a greater awareness of diet and exercise, with support from staff and an improved physical health. Participants will be encouraged to monitor their food, activity and sleep (FAS diary), which will increase their awareness of a healthy lifestyle and the benefits thereof. The majority of outcome measures will be routine measures (BMI, blood pressure) and there will be three additional questionnaires administered every three months, each taking approximately ten minutes. The patients will also undergo questionnaires to assess their attitude towards the study (qualitative research) prior to the start of the study, at 12 months and upon completion of the study. This will be should take up to 15 minutes. These will be carried out at the patient's own convenience. Additionally, the patient will be asked to wear an activity monitor (in the form of a watch) for one week every three months. This has been used in previous exercise- based studies at St Andrew's and they have been shown to be well tolerated and the patients are interested to understand the amount of activity that they undergo on a daily basis. .

Confidentiality:

All of the data collected during the study will stored in a password-protected file on the St Andrew's server and only available to names members of the research team. This is highlighted in the patient information sheet.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 35.0 kg/m2 or above or BMI of 32.5 kg/m2 for people from South Asian, Chinese, other Asian, Middle Eastern, Black African or African-Caribbean family
* Aged 18 or above
* Able to give informed consent, as assessed by their RC. In the context of participation in this trial 'informed' consent includes having an understanding of the dietary and exercises changes needed for the treatment to be effective
* Currently prescribed olanzapine or clozapine
* Currently in an inpatient service
* Sufficient level of English to read and understand the information sheet (may require verbal explanation from support from staff)

Exclusion Criteria:

* Aged 17 or under
* Meet any of the contraindications, including hypersensitivity to the active substance or to any of the excipients
* Pregnant or likely to become pregnant
* Diagnoses of dementia or Huntington's disease
* On a PICU/acute ward
* Discharge anticipated to be in 6 months' time or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Weight | 36 months
  This will be calculated in kg and the patient weighed on a weekly basis. This will be calculated for the 12 months prior to enrolment into the trial according to the patient's clinical notes and on a weekly basis during the 24 months of the trial.
Body mass index | 36 months
  The BMI will be calculated according to the ratio of body mass (kg) and height (cm) and will be measured on a weekly basis. This will be calculated for the 12 months prior to enrolment into the trial according to the patient's clinical notes and on a weekly basis during the 24 months of the trial
Waist circumference | 36 months
  Waist circumference will be measured in cm. This will be calculated for the 12 months prior to enrolment into the trial according to the patient's clinical notes and on a weekly basis during the 24 months of the trial.
Blood pressure | 36 months
  This will be calculated in mm Hg as both systolic and diastolic blood pressure. This will be calculated for the 12 months prior to enrolment into the trial according to the patient's clinical notes and on a weekly basis during the 24 months of the trial. It will be measured while the patient is in a sitting state.
Heart rate | 36 months
  This will be calculated as beats per minute and will be measured over a 30 second time period. This will be calculated for the 12 months prior to enrolment into the trial according to the patient's clinical notes and on a weekly basis during the 24 months of the trial.

SECONDARY OUTCOMES:
To explore the potential relationship between patient adherence to STEP@STAH and changes in quality of life | 24 months
  Variables will be assessed to understand the mechanism by which the therapy has influenced the patient's overall lifestyle and contributed to changes in their physical health. Specifically, we aim to determine whether the STEP@STAH therapy has affected their:
  - Quality of life
  To do this, the following additional outcome measures will be collected and correlated with the physical outcomes:
  • IWQOL Lite CT Health Survey This will be measured at baseline and then every three months over the course of the trial
To explore the potential relationship between patient adherence to STEP@STAH and changes in wellbeing | 24 months
  Variables will be assessed to understand the mechanism by which the therapy has influenced the patient's overall lifestyle and contributed to changes in their physical health. Specifically, we aim to determine whether the STEP@STAH therapy has affected their:
  - Appetite
  To do this, the following additional outcome measures will be collected and correlated with the physical outcomes:
  • Control of Eating Questionnaire (CoEQ) This will be measured at baseline and at weeks 8, 16, 28 & 56, 78, 104.
To explore the potential relationship between patient adherence to STEP@STAH and changes in wellbeing | 24 months
  Variables will be assessed to understand the mechanism by which the therapy has influenced the patient's overall lifestyle and contributed to changes in their physical health. Specifically, we aim to determine whether the STEP@STAH therapy has affected their:
  - Appetite
  To do this, the following additional outcome measures will be collected and correlated with the physical outcomes:
  • Leeds Food Preference Questionnaire (LFPQ) This will be measured at baseline and then every six months thereafter.
To explore the potential relationship between patient adherence to STEP@STAH and changes in physical activity | 24 months
  Variables will be assessed to understand the mechanism by which the therapy has influenced the patient's overall lifestyle and contributed to changes in their physical health. Specifically, we aim to determine whether the STEP@STAH therapy has affected their level of physical activity & exercise. Patients will wear an ActiGraph activity monitor to measure their physical activity (step count) for 1 week every quarter starting 3 months after enrolment.
To explore the potential relationship between co-morbidities and impact of STEP@STAH | 24 months
  All patients will be monitored for physical health problems, particularly type 2 diabetes for which semaglutide has been prescribed. Their medical history will be assessed upon completion of the study to determine whether any incidents of note, such as the development of critical physical health incidents, has occurred and whether these could be attributed to their participation in the current trial
To qualitatively explore the barriers, facilitators and acceptability of the intervention from both patient and staff perspectives | 24 months
  Transcripts will be coded using thematic analysis methods. Initial codes will be generated from the transcripts to capture meaningful units of data related to barriers, facilitators, and acceptability. Codes will be organised into broader themes and sub-themes through iterative review and comparison. Themes will represent patterns and recurring topics across the data. Themes will be interpreted in relation to the research questions, aiming to provide insights into factors influencing the intervention's implementation and acceptance among patients and staff

CONTACTS AND LOCATIONS:
Overall Officials: Kieran C Breen, PhD, Principal Investigator — St Andrew's Healthcare
Locations (1):
- St Andrew's Healthcare, Northampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised physical healthcare data on clinical outcomes will be available upon request upon completion of the study
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The IPD will be available upon completion of he trial for a period of up to three years after publication of the trial results.
Access Criteria: All requests will be considered by the trial steering group.